CLINICAL TRIAL: NCT00040170
Title: Randomized Multicenter Phase II Study Evaluating Two Dosing Schedules of TG4010(MVA-MUC1-IL2) in Patients With Adenocarcinoma of the Prostate
Brief Title: Vaccine Study of MVA-MUC1-IL2 in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Transgene (Industry)
Collaborators: University of California, Los Angeles (Other); The Cleveland Clinic (Other); University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG4010.03; NCT00040976 (obsolete NCT alias)
Record Dates: First submitted 2002-06-21; First posted 2002-06-25 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2006-10

CONDITIONS: Prostatic Neoplasms
Keywords: Adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: MVA-MUC1-IL2

SUMMARY:
This study involves the use of an experimental product, TG4010. The purpose of the study is to determine if TG4010 can stimulate the body's immune system to help it fight the cancer.

DETAILED DESCRIPTION:
The experimental product, TG4010, is a modified vaccinia virus (already used in humans) into which two (2) genes have been placed. One gene is for a protein (MUC1) found in cancer cells. The second gene is for human interleukin 2 (IL2) which the body's immune system makes to help it fight cancer. The TG4010 is given as an injection under the skin (subcutaneous) once a week for six weeks followed by a schedule of every three weeks or every three weeks for the first twelve (12) weeks. If the therapy is working, it can be continued for up to 9 months until no further improvement or until the patient gets worse for as long as it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Rising PSA after surgery or radiation for prostate cancer

Exclusion Criteria:

* Metastasis or local disease
* Prior hormone treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA, Los Angeles, California
  - Cleveland Clinic Foundation, Cleveland, Ohio